CLINICAL TRIAL: NCT02197923
Title: Norwegian Adenomyosis Study: Pathophysiology, Peristalsis, Expression Profiling and Diagnosis, Part 2
Brief Title: Norwegian Adenomyosis Study II: Gene Expression Profiling of Adenomyosis
Acronym: NAPPED II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Tina Tellum, MD, Oslo University Hospital
Other Study IDs: 2014/637b
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Adenomyosis
Keywords: Menorrhagia; Dysmenorrhea; Pelvic pain; expression profiling; uterine biopsies; serum hormones
MeSH Terms: conditions — Adenomyosis; Menorrhagia; Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and biopsies from uterine myometria and uterine endometria
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Biopsy: adenomyosis: Myometrial biopsy Pipelle
  Interventions: Procedure: Myometrial biopsy; Procedure: endometrial biopsy
- Biopsy: Healthy: Myometrial Biopsy Pipelle
  Interventions: Procedure: Myometrial biopsy; Procedure: endometrial biopsy

INTERVENTIONS:
Procedure: Myometrial biopsy — transvaginal ultrasound guided biopsy of the myometria
Procedure: endometrial biopsy — transcervical endometrial biopsy
  Other Names: Pipelle

SUMMARY:
Adenomyosis is characterized by the appearance of endometrial cells in the muscular layer of the uterus. It affects about 15-20% of the female population.

The symptoms of adenomyosis are heavy menstrual bleedings and painful menstruation (dysmenorrhea) and in addition chronic pelvic pain. Subfertility and infertility have been correlated with adenomyosis.

Parity, age and uterine abrasion increase the risk of adenomyosis. Hormonal factors such as local hyperestrogenism and elevated levels of prolactin (PRL) have been identified, but autoimmune and mechanical factors are also hypothesized.

Regarding treatment, the most effective measure is hysterectomy. As this is a very drastic measure in younger women, levonogestrel-releasing intrauterine devices, Gonadotropin releasing hormone (GnRH)-analogues, Danazol, uterine embolization and endometrial ablation have been tried, but studies are few in number, retrospective, and have small sample sizes.

Adenomyosis has so far not been subject to extensive research efforts. The pathogenesis of adenomyosis remains still unclear, there are not many satisfying treatment options and diagnostics include mostly magnetic resonance imaging (MRI) and histology.

The investigators designed a series of 3 studies with a broad approach in understanding adenomyosis. This is part 2.

In this study the investigators take both tissue samples and blood samples that will be investigated in order to understand the basic processes leading to adenomyosis.

DETAILED DESCRIPTION:
Biopsy of focal adenomyosis of the myometrium:

This will be an extension of the NAPPED1-study. The investigators will perform ultrasound-guided transvaginal biopsies of the myometrium and collect venous blood samples.

As recent studies have suggested abnormalities in the regulation of specific genes in the development of adenomyosis, the investigators want to investigate differentially expressed genes in adenomyosis compared to eutopic endometrium. Using microarrays, the investigators can simultaneously screen differences in expression of thousands of genes in samples from the two groups. Profiling studies performed on endometrium of healthy individuals and of endometriosis show results that enable identification of biological processes and molecular mechanisms. Expression profiles can be used to identify molecular targets for therapeutic purposes. There are some very interesting studies that investigate drug treatment on a molecular level e.g. the effect of Danazol treatment on eutopic and ectopic endometrial tissue, but intramural adenomyosis has not been subject to gene profiling yet.

Tissue samples can be easily obtained after hysterectomy, but those samples will only represent older women, and cannot be used for consecutive monitoring of biochemical effects of treatment, as the uterus is removed. In order to investigate the pathophysiology of adenomyosis in younger women, and compare it to those in older individuals, as well as to evaluate effects of treatment, it is necessary to be able to obtain in-vivo samples.

The plan is therefore to take transvaginal, ultrasound-guided biopsy-samples from the uterus (myometrium) of all included patients at the beginning of their surgery, when the patient is under full anesthesia. The safety of comparable procedures has been shown in prior studies, but the investigators will further validate the safety of this method. The investigators believe that an in-vivo biopsy is a safe measure, and that representative samples of adenomyosis can be obtained.

The challenge with adenomyosis is that it is located intramyometrially. A transcervical biopsy will contaminate the sample with eutopic endometria, therefore it is most meaningful to take the biopsy transvaginally, but not through the cavity. After obtaining the biopsy sample, it will be examined histologically by imprint, to confirm if glandular cells are contained where expected. When good routines show a reliable level of specificity, the investigators will go further by selecting approximately 10 patients for gene profiling of adenomyosis. The investigators will also use endometrial biopsies (Pipelle) from those patients to see if there is a difference between intramural adenomyosis and their eutopic endometria. Most patients that undergo hysterectomy have taken a pipelle-biopsy routinely.

The levels of prolactin, Anti-müllerian hormone (AMH), Follicle stimulating hormone (FSH), luteinizing hormone (LH) and estrogen will also be taken, in order to determine if the severity of adenomyosis is only related to age as shown before, or also to hormonal activity.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal women aged 30 - 50 years old scheduled for vaginal, abdominal or laparoscopic total hysterectomy one or more of the following clinical symptoms:

* bleeding disorders (menorrhagia, irregular bleeding, hypermenorrhoea),
* chronic pelvic pain,
* dysmenorrhoea,
* or dyspareunia junction zone definable

Exclusion Criteria:

* postmenopausal women,
* pregnancy
* gynecological cancer
* GnRH analog therapy or systemic hormone therapy in the last three months prior to hysterectomy
* junctional zone not identifiable

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women referred to our clinic and volunteering to participate
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-08-06 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of biopsies for adenomyotic tissue in percent (%) | At time of hysterectomy
  Sensitivity and specificity of ultrasound guided myometrial biopsies for adenomyotic tissue

SECONDARY OUTCOMES:
multiple comparison of gene expression, measured in fold | at time of biopsy taking
  Expression profile for proliferative and invasive genes in adenomyotic tissue and surrounding stromal cells compared to healthy individuals, in fold
Frequency of complications related to biopsy taking in percent (%) | through 1 hour after biopsytaking
Serum levels of prolactin in mU/L | at time of hysterectomy
  Serum levels of prolactin
Serum level of ER, in nmol/L | at time of hysterectomy
  Serum level of estrogen.
Serum levels of FSH in U/L | at time of hysterectomy
  Levels of follicle stimulating hormone.
Serum levels of AMH in pmol/L | at time of hysterectomy
  Levels of Anti-Mullerian hormone.
Serum levels of LH in U/L | at time of hysterectomy
  Levels of luteinizing hormone.
difference hormone serum-levels in fold | at time of hysterectomy
  Comparison of serum-levels of PRL, FSH, AMH, LH and ER in patients with and without adenomyosis

CONTACTS AND LOCATIONS:
Overall Officials: Erik Qvigstad, PhD, MD, Study Chair — Oslo University Hospital, Ullevål; Tina Tellum, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Gynecological department, Oslo University Hospital, Ullevål, Oslo, Norway